CLINICAL TRIAL: NCT05620368
Title: Mindfulness-Based Online Support Program for Mothers of Children With Disabilities
Brief Title: Mindfulness for Mothers of Children With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: University of Silesia in Katowice (Unknown); Jan Dlugosz University in Czestochowa (Other)
Responsible Party: Principal Investigator, Błażej Cieślik, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01/2021
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-12

CONDITIONS: Parental Burnout; Caregiver Burnout
Keywords: parental burnout; meditation; mindfulness; self-compassion; stress level; parents of children with disability; autism; quality of life
MeSH Terms: conditions — Caregiver Burden; Autistic Disorder | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based teleintervention (Experimental): 8-week Mindfulness and Compassionate Living Course (MCLC). The course will be held online (using the Zoom platform) with weekly sessions lasting 2.5 hours each, as well as a day of silent practice (mini-retreat of 4 hours).
  Interventions: Behavioral: Mindfulness and Compassionate Living Course (MCLC)
- Usual care intervention (Active Comparator): The facility provides psychological support for parents as needed and at the request of the parent. Support includes individual support of a psychologist (1h / week), consultation with a teacher (special pedagogue and early school education teacher, 1h / week), individual consultation with observation of a child with a Venetian mirror (1h / week).
  Interventions: Behavioral: Usual care intervention

INTERVENTIONS:
Behavioral: Mindfulness and Compassionate Living Course (MCLC) — The course will be held online (using the Zoom platform) with weekly sessions lasting 2.5 hours each, as well as a day of silent practice (mini-retreat of 4 hours) between sessions 6 and 7.
  On the structural level, every course session consists of four elements: (1) an educational input, (2) mindfulness and compassion exercises (eg, sitting meditation, body scan, mindful walking, self-compassion break), (3) a reflection of one's practice (inquiry), (4) and home assignments.
  Arms: Mindfulness-based teleintervention
Behavioral: Usual care intervention — If necessary, psychological support is organized at the request of the parent.
  Support includes individual support of a psychologist (1h / week), consultation with a teacher (special pedagogue and early school education teacher, 1h / week), individual consultation with observation of a child with a Venetian mirror (1h / week).
  Arms: Usual care intervention

SUMMARY:
The main objective of this study is to evaluate the effectiveness of an eight-week mindfulness-based teleintervention in improving quality of life, parental burnout, self-compassion, and stress level in mothers of children with disabilities.

DETAILED DESCRIPTION:
Parenthood is accompanied by significant mental and physical effort accompanied by different sources of long-term stress and encumbrance. The results of this research indicate serious difficulties in the functioning of parents of children with disabilities, such as pain, emotional and physical discomfort, anxiety, depression, and problems resulting from the realization of everyday life activities combined with the care of the child. They indicate how serious this crisis is and how important life constraints it brings to the individual and the social functioning of the family.

A parent's ability to adapt to stressful situations depends on several variables, including an individual's psychological strengths, individual and family resources, and the type of coping strategies utilized. Parental burnout is defined as a syndrome that occurs in response to chronic parental stress. The risk of parental burnout is related to family functioning. In the concept of family as an interactional system, "family adaptability is the degree to which the family is flexible and can regain equilibrium in stressful and challenging situations or environments".

Positive coping styles such as positive perceptions and effective problem-solving skills were associated with successful family adaptation and resilience. Twenty years ago, the concept of mindful parenting was introduced as an alternative to traditional discipline-oriented methods by focusing on the quality of a parent's presence in the parent-child dyad. It focuses on cultivating mindfulness and attunement with the parent's inner experience while interacting with the child, and feeling the full range of emotions related to parenting. Mindful parenting involves cultivating non-judgmental awareness of the unfolding of internal and external experiences in daily life, practicing emotion regulation skills, learning about adaptive responses to distress, and developing a self-compassionate attitude toward one's fallibility, limitations, and suffering.

Compassion- and mindfulness-based interventions (CMBIs) hold promise in supporting parental resilience by enabling adaptive stress appraisal and coping, mindful parenting, and self-compassion. These interventions also aimed to reduce social isolation by increasing the capacity for connections. Perceived social support, an aspect of compassionate behavior, is a potent buffer against stress on health outcomes.

Therefore, the main objective of this study is to evaluate the effectiveness of an eight-week mindfulness-based teleintervention in improving quality of life, parental burnout, self-compassion, and stress level in mothers of children with disabilities. The investigators hypothesize that the mindfulness-based teleintervention compared with the control group will lead to (A) an improvement in positive aspects of mental health, including quality of life, and self-compassion, and (B) a reduction in psychopathological variables including perceived stress and parental burnout.

ELIGIBILITY:
Inclusion Criteria:

* mother of childern with disabilities

Exclusion Criteria:

* substance abuse;
* participation in another therapeutic project or individual psychotherapy;
* antidepressant treatment.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Families in Early Intervention Quality of Life (FEIQoL) | 15 minutes
  Families in Early Intervention Quality of Life (FEIQoL) questionnaire will be used for assessing the quality of life. Participants answer 40 items using a five-point Likert scale (1, 'poor' to 5, 'excellent') in the aspects of family life (24 items), and child's functioning (16 items).

SECONDARY OUTCOMES:
Parental Burnout Measure (PBM-12) | 7 minutes
  Parental Burnout will be assessed with the Parental Burnout Measure (PBM-12) measures parental burnout in two dimensions: exhaustion and helplessness. Both dimensions are measured as a sum of 6 items, answered on a 4-point Likert scale (1, 'never' to 4, 'very often'). Fully satisfactory internal reliability indicators (Cronbach's alpha) were reached by all burnout measures - PBM-12 total score (.90), exhaustion subscale (.88), and helplessness sub-scale (.80).
Self-Compassion Scale (SCS) | 7 minutes
  To assess self-compassion we will use a polish adaptation of the Self-Compassion Scale (SCS). Items on the SCS use a five-point Likert scale to measure conformity (1, 'almost never' to 5, 'almost always'). The final SCS score ranges from 26 to 130. A higher score indicates a higher level of self-compassion. This scale has good internal consistency and test-retest reliability (.93).
Perceived Stress Scale (PSS-10) | 7 minutes
  The 10-item Perceived Stress Scale (PSS-10) will be used to measure self-reported stress. This scale includes 10 questions, with answers ranked using a 5-point Likert scale, and assesses stressful experiences and responses to stress over the previous 4 weeks. Scores range from 0 to 56, with higher scores indicating higher levels of perceived stress.
Ego Resilience Scale (ER89) | 7 minutes
  The Ego-Resiliency Scale (ER89) measures the construct of ego-resiliency, which refers to the dynamic capacity of an individual to modify a characteristic level of ego-control, in either direction, as a function of the demand characteristics of the environmental context, so as to preserve or enhance system equilibration. It consists of 14 items, each responded to on a 4-point scale (1 = "does not apply at all"; 2 = "applies slightly, if at all"; 3 = "applies somewhat"; and 4 = "applies very strongly").

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Sekułowicz, Professor, Study Chair — Wroclaw University of Health and Sport Sciences; Krystyna Boroń-Krupińska, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences; Sylwia Wrona, PhD, Principal Investigator — University of Silesia in Katowice
Locations (3):
- Poland (3):
  - Wroclaw University of Health and Sport Sciences, Wroclaw, Lower Silesian Voivodeship
  - Jan Dlugosz University in Czestochowa, Częstochowa, Upper Silesia
  - University of Silesia in Katowice, Katowice, Upper Silesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zessin U, Dickhauser O, Garbade S. The Relationship Between Self-Compassion and Well-Being: A Meta-Analysis. Appl Psychol Health Well Being. 2015 Nov;7(3):340-64. doi: 10.1111/aphw.12051. Epub 2015 Aug 26. PMID 26311196
- [Background] Allen AB, Leary MR. Self-Compassion, Stress, and Coping. Soc Personal Psychol Compass. 2010 Feb 1;4(2):107-118. doi: 10.1111/j.1751-9004.2009.00246.x. PMID 20686629
- [Background] Neece CL, Chan N, Klein K, Roberts L, Fenning RM. Mindfulness-Based Stress Reduction for Parents of Children with Developmental Delays: Understanding the Experiences of Latino Families. Mindfulness (N Y). 2019 Jun;10(6):1017-1030. doi: 10.1007/s12671-018-1011-3. Epub 2018 Sep 6. PMID 31191735
- [Background] Bohadana G, Morrissey S, Paynter J. Self-compassion: A Novel Predictor of Stress and Quality of Life in Parents of Children with Autism Spectrum Disorder. J Autism Dev Disord. 2019 Oct;49(10):4039-4052. doi: 10.1007/s10803-019-04121-x. PMID 31267283
- [Background] Bohadana G, Morrissey S, Paynter J. Self-Compassion in Mothers of Children with Autism Spectrum Disorder: A Qualitative Analysis. J Autism Dev Disord. 2021 Apr;51(4):1290-1303. doi: 10.1007/s10803-020-04612-2. PMID 32656737
- [Background] Bogels SM, Lehtonen A, Restifo K. Mindful Parenting in Mental Health Care. Mindfulness (N Y). 2010 Jun;1(2):107-120. doi: 10.1007/s12671-010-0014-5. Epub 2010 May 25. PMID 21125026
- [Background] Wang H, Wang Q, Hu X, Han ZR. Mindfulness and Stress Among Parents of Children with Autism Spectrum Disorder in China. J Autism Dev Disord. 2022 May;52(5):2035-2045. doi: 10.1007/s10803-021-05011-x. Epub 2021 May 29. PMID 34050845
- [Background] Cousineau TM, Hobbs LM, Arthur KC. The Role of Compassion and Mindfulness in Building Parental Resilience When Caring for Children With Chronic Conditions: A Conceptual Model. Front Psychol. 2019 Aug 5;10:1602. doi: 10.3389/fpsyg.2019.01602. eCollection 2019. PMID 31428005
- [Background] Duncan LG, Coatsworth JD, Greenberg MT. A model of mindful parenting: implications for parent-child relationships and prevention research. Clin Child Fam Psychol Rev. 2009 Sep;12(3):255-70. doi: 10.1007/s10567-009-0046-3. PMID 19412664
- [Background] Ettman CK, Abdalla SM, Cohen GH, Sampson L, Vivier PM, Galea S. Prevalence of Depression Symptoms in US Adults Before and During the COVID-19 Pandemic. JAMA Netw Open. 2020 Sep 1;3(9):e2019686. doi: 10.1001/jamanetworkopen.2020.19686. PMID 32876685
- [Background] Friis AM, Johnson MH, Cutfield RG, Consedine NS. Kindness Matters: A Randomized Controlled Trial of a Mindful Self-Compassion Intervention Improves Depression, Distress, and HbA1c Among Patients With Diabetes. Diabetes Care. 2016 Nov;39(11):1963-1971. doi: 10.2337/dc16-0416. Epub 2016 Jun 22. PMID 27335319
- [Background] Homan KJ, Sirois FM. Self-compassion and physical health: Exploring the roles of perceived stress and health-promoting behaviors. Health Psychol Open. 2017 Sep 14;4(2):2055102917729542. doi: 10.1177/2055102917729542. eCollection 2017 Jul-Dec. PMID 29379620
- [Background] Ten Hoopen LW, de Nijs PFA, Duvekot J, Greaves-Lord K, Hillegers MHJ, Brouwer WBF, Hakkaart-van Roijen L. Children with an Autism Spectrum Disorder and Their Caregivers: Capturing Health-Related and Care-Related Quality of Life. J Autism Dev Disord. 2020 Jan;50(1):263-277. doi: 10.1007/s10803-019-04249-w. PMID 31625009
- [Background] Kuhlthau KA, Luberto CM, Traeger L, Millstein RA, Perez GK, Lindly OJ, Chad-Friedman E, Proszynski J, Park ER. A Virtual Resiliency Intervention for Parents of Children with Autism: A Randomized Pilot Trial. J Autism Dev Disord. 2020 Jul;50(7):2513-2526. doi: 10.1007/s10803-019-03976-4. PMID 30900195
- [Background] Robinson S, Hastings RP, Weiss JA, Pagavathsing J, Lunsky Y. Self-compassion and psychological distress in parents of young people and adults with intellectual and developmental disabilities. J Appl Res Intellect Disabil. 2018 May;31(3):454-458. doi: 10.1111/jar.12423. Epub 2017 Nov 9. PMID 29119672
- [Background] Turnage D, Conner N. Quality of life of parents of children with Autism Spectrum Disorder: An integrative literature review. J Spec Pediatr Nurs. 2022 Oct;27(4):e12391. doi: 10.1111/jspn.12391. Epub 2022 Aug 20. PMID 35986656